CLINICAL TRIAL: NCT01691287
Title: MICHAEL Method- Fulfilling Individual Potential to Attain Excellence - as a Tool for Improving Metabolic Control and Quality of Life Among Adolescence With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: rmc006444ctil
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Metabolic Control; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Michael Method (Experimental): 14 group meeting, taking place once a week during 14 consecutive weeks
  Interventions: Behavioral: Michael Method

INTERVENTIONS:
Behavioral: Michael Method

SUMMARY:
Type 1 diabetes is the most common childhood disease. Treatment of diabetes requires personal checks of blood sugar levels, injecting insulin, changing eating habits and physical exercise, which requires a real change in the life of the child & adolescent and can cause significant damage to the quality of life as well.

Compliance to treatment is a major challenge for all patients and mostly to adolescence, which often worsen their diabetes control at that age.

The Michael Method is a unique, holistic program to develop and realize an individual's emotional, intellectual and behavioral potential, which is based on the belief that every human being can excel in every field they choose. The method was developed in 1988 by a multi-disciplinary team of professional academic in Israel. Today the Israeli education system implements the method in Junior High Schools and High Schools in diverse educational sectors. The program is taught at many other various frameworks: teachers' continuing education programs, colleges, programs run by the Ministries of Defense and Social Welfare, the National Insurance Institute, the National Electric Corporation and in many other public and private frameworks.

The proposed study is aimed to assess whether the Michael Method can be used as a tool for improving metabolic control and quality of life among uncontrolled adolescence with type 1 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes at least 1 year prior to study inclusion
* 12-17 years old
* HbA1c > 7.8%

Exclusion Criteria:

- Incapability to comply with all study requirements

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Metabolic Control measured as HbA1c level | at the end of the study - after 15 weeks

SECONDARY OUTCOMES:
Diabetes Quality of Life questionnaire (DQOLY) | At the end of the study- after 15 weeks
Self assessment questionnaire | At the end of the study- after 15 weeks
Number of severe hypoglycemic events | at the end of the study-after 15 weeks
Number of Diabetic Keto Acidosis events | at the end of the study- after 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Medical Center, Petah-TTikva, Israel